CLINICAL TRIAL: NCT05040321
Title: A Proof of Concept Trial of a Sirtuin-NAD Activator in Alzheimer's Disease
Brief Title: Sirtuin-NAD Activator in Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P001366; MIB-AD (Other: Metro International Biotech, LLC)
Record Dates: First submitted 2021-07-27; First posted 2021-09-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer's Disease (Incl Subtypes); Dementia
Keywords: Dementia; NAD; MIB-626
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: We will use an IRB approved structured telephone screen to ask about basic demographics, major study required inclusion/exclusion criteria, and questions regarding MR contraindications. Those who do not have major exclusionary conditions identified during the telephone screening and who are interested in participating will be invited for an in-person visit. During the in-person screening visit, informed consent will be obtained, and subjects will undergo screening neuropsychological testing and medical evaluation.
  Subjects will come back after their initial screening visit for 2 more screening visits before they are found eligible and go through Baseline visits, also known as Day 0. Subjects will receive MIB-626 or placebo twice a day for 90 days. There will be one more visit, known as the washout period, at day 105. The total completion of all of the study visits will be 8 visits, for 150 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind; the participants, care provider, investigators and outcome assessors are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIB-626 (Experimental): Subjects will either take MIB-626 or placebo tablet twice a day for 90 days. For those who receive MIB-626, we plan on giving subjects 1000mg of the drug, twice a day for 90 days. MIB-626 will be in two 500mg tablets.
  Interventions: Drug: MIB-626
- Placebo Tablet (Placebo Comparator): Subjects will be randomized to receive either the placebo or MIB-626 tablets twice a day orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIB-626 — Participants will be randomized to either receive MIB-626 or matching placebo. The proposed intervention - targets multiple contributors to the pathology of AD; MIB-626 improves mitochondrial function, bioenergetics, and insulin sensitivity, inhibits A beta accumulation by reducing its synthesis and increasing its clearance, reduces neuroinflammation, exerts neuronal protective effects, and promotes neuronal regeneration and connectivity in preclinical models.
  Arms: MIB-626
Drug: Placebo — Subjects will be randomized to receive either the placebo or 1000 mg MIB-626 twice daily orally.
  Arms: Placebo Tablet

SUMMARY:
The primary objectives are to:

1. To determine whether MIB-626, after its daily oral administration, penetrates the blood-brain barrier in humans by measuring the cerebrospinal fluid (CSF) concentrations of MIB-626 and its key metabolites, nicotinamide (NAM), NR, 2-PY, and MeNAM at baseline and on day 90 at steady state.
2. To evaluate whether oral MIB-626 administration engages the sirtuin-NAD pathway by determining the abundance of NAD (a SIRT1 substrate) in the brain using ultra-high field 7T magnetic resonance spectroscopy and in peripheral blood mononuclear cells using a validated LC-MS/MS assay.
3. To determine whether MIB-626 alters the circulating biomarkers of aging that the geroscience experts have recommended (HbA1C, IGF1, T3, IL6, TNF, and urinary F2-isoprostane).

DETAILED DESCRIPTION:
The sirtuin family of nicotinamide adenine dinucleotide (NAD)-dependent deacetylase enzymes are important regulators of the aging process and mediate many of the beneficial effects of caloric restriction. The upregulation of the sirtuin-NAD pathway by increasing intracellular NAD through administration of NAD precursors, such as niacinamide β nicotinamide mononucleotide (βNMN) and nicotinamide riboside, has been shown to engage fundamental mechanisms of aging and prevent or attenuate Alzheimer's disease (AD) pathology in preclinical models. In contrast to many AD drugs in development that target one mechanism, NAD precursors may prevent AD pathology by multiple mechanisms: by improving mitochondrial energetics; inducing a switch to non-amyloidogenic processing of amyloid precursor protein (APP) due to increased α-secretase activity; reducing the synthesis of oligomerized Aβ peptides; preventing microglia-dependent Aβ toxicity; attenuating neuroinflammation; promoting neuronal regeneration; and improving insulin action.

In spite of the promising preclinical data, the human studies of the clinical pharmacology, physiologic effects, efficacy, and safety of NAD precursors have been few and constrained by several methodological barriers. First, βNMN and nicotinamide riboside (NR) are sold as dietary supplements and these over-the-counter products have suffered from variable manufacturing quality. Second, there is only limited information available on the pharmacokinetics (PK) and pharmacodynamics (PD) of βNMN and NR in humans, and the doses used in some initial studies were low. Third, NAD and many other metabolites of βNMN and NR are labile and susceptible to rapid degradation ex vivo. Furthermore, the assays for the measurement of intracellular NAD, βNMN, and its metabolites have been challenging. Although NR and βNMN have been shown to cross the blood-brain barrier, attenuate AD pathology, and improve cognitive function in preclinical models, no clinical trials have been conducted to determine whether βNMN crosses the blood-brain barrier or engages the target mechanisms in humans.

To overcome these methodological barriers, we have characterized the pharmacokinetics of MIB-626 in phase 1 studies, validated the methods for measuring intracellular NAD, and established the procedures for blood collection to ensure pre-analytical stability. These phase 1 studies have shown that a regimen of 1 g MIB-626 twice daily is safe and effective in substantially raising circulating NAD levels in healthy adults (preliminary data). These foundational methods and single and multiple-dose pharmacokinetic studies have paved the way for the proposed 90-day randomized trial in 24 mild AD dementia participants to determine whether MIB-626 crosses the blood-brain barrier, engages the hypothesized target mechanism, and whether it improves the biomarkers of aging. We hypothesize that MIB-626 administration at the proposed dose will cross the blood-brain barrier and be associated with an increase in brain NAD. Because of the important role of the sirtuin-NAD pathway in regulation of the mechanisms of aging, we will also assess whether MIB-626 is more efficacious than placebo in improving biomarkers of aging in participants with mild AD dementia.

ELIGIBILITY:
Inclusion Criteria:

1. A man or a woman between the ages of 55 and 85 years (inclusive)
2. Meets National Institute on Aging-Alzheimer's Association (NIA-AA) clinical diagnostic criteria for AD dementia
3. Has evidence of AD pathological process by a positive amyloid assessment with cerebrospinal fluid (CSF) Aβ42
4. Has a Clinical Dementia Rating (CDR) global score of 0.5 or 1
5. Has a Mini-Mental State Exam (MMSE) Score of 18 to 26 (inclusive)
6. Has a 15-item Geriatric Depression Scale (GDS) score of < 6
7. Impaired memory performance below education adjusted cut-off score on the Logical Memory II subscale delayed paragraph recall (LM-IIa) of the Wechsler Memory Scale-Revised (WMS-R) (≥16 years: ≤8; 8-15 years: ≤4; 0-7 years: ≤2)
8. May take Food and Drug Administration (FDA) approved medications for the treatment of AD dementia (cholinesterase inhibitors and/or memantine), but if taking such medications, they must be stable for at least 8 weeks before screening
9. Has adequate visual and auditory acuity to participate in neuropsychological testing and other study assessments
10. Has the availability of an informant (study partner) who has regular contact with the participant and knows him/her well
11. Is willing and able to participate in all assessments in English
12. Is capable of providing written informed consent

Exclusion Criteria:

Subjects may not be enrolled if:

1. Neurologic diseases: Any significant neurologic disease other than AD that can lead to cognitive impairment, such as Parkinson's disease, vascular dementia, dementia with Lewy bodies, frontotemporal dementia, Huntington's disease, normal pressure hydrocephalus, corticobasal syndrome, brain tumor, seizure disorder, subdural hematoma (within the last 1 year), multiple sclerosis, or history of significant head trauma (e.g. loss of consciousness for 30 minutes or more) followed by persistent neurologic deficits or known structural brain abnormalities.
2. Neuroimaging: Baseline or prior magnetic resonance imaging (MRI) scans with evidence of cortical stroke or hemorrhage, strategically located lacunar stroke (ex: left thalamus), or severe small vessel ischemic disease.
3. History of alcohol or substance use disorder or dependence (DSM V criteria) within the last 2 years.
4. Psychiatric disorder: Major depressive disorder (within the last 1 year), bipolar disorder, schizophrenia (DSM V criteria), or current major psychotic symptoms or behavioral problems that could interfere with study procedures.
5. Any significant systemic illness or unstable medical condition, which could obfuscate cognitive aging or neurodegenerative trajectories or affect valid cognitive and self-report measurements.
6. Excluded medications: Niacin or dietary supplements containing nicotinamide mononucleotide (NMN) or nicotinamide riboside (NR); antipsychotic medications, antidepressant medications with anticholinergic side effects. Washout from psychoactive medications for at least 8 weeks before screening.
7. Current use of anticoagulants; significant back or spine disease that would make a lumbar puncture difficult or unsafe as determined by a clinician.
8. Other laboratory abnormalities: Has AST or ALT > 3 times the upper limit of normal; serum creatinine > 2.0 mg/d; HbA1C > 8.5%
9. Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months or 5 half-lives, whichever is shorter
10. Other medical conditions which, in the opinion of the investigator, would jeopardize safety or impact the validity of the study results.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in CSF concentrations of MIB-626 | 90 days
  change in CSF concentrations of MIB-626 at baseline and on day 90 at steady state

SECONDARY OUTCOMES:
change in CSF concentrations of MIB-626 metabolites, nicotinamide (NAM), NR, 2-PY, and MeNAM | 90 days
  change from baseline to day 90 in CSF concentrations of MIB-626 metabolites NAM, NR, 2-PY and MeNAM
  The concentrations of MIB-626's metabolites NAM, NR, 2-PY, and MeNAM will be measured in the CSF
change in the abundance of NAD in the brain using ultra-high field 7T magnetic resonance spectroscopy | 90 days
  change from baseline to day 90 in the abundance of NAD in the brain using ultra-high field 7T magnetic resonance spectroscopy
change in NAD concentrations in peripheral blood mononuclear cells | 90 days
  change from baseline to day 90 in NAD concentrations in peripheral blood mononuclear cells using validated LC-MS/MS assay
change in the concentration of biomarkers of aging recommended (HbA1C, IGF1, T3, IL6, TNF-alpha, and urinary F2-isoprostane) | 90 days
  change from baseline to day 90 in the concentration of biomarkers of aging recommended (HbA1C, IGF1, T3, IL6, TNF-alpha, and urinary F2-isoprostane)

OTHER OUTCOMES:
change in CSF concentrations of biomarkers of amyloid deposition (Aβ-42, Aβ-40), neuronal/axonal degeneration (t-tau, p-tau, NFL), synaptic function (neurogranin) and neuroinflammation (YKL40, GFAP) | 90 days
  change from baseline to day 90 in CSF concentrations of biomarkers of amyloid deposition (Aβ-42, Aβ-40).
Change in circulating biomarkers of amyloid deposition (Aβ-42, Aβ-40), neuronal/axonal degeneration (t-tau, p-tau, NFL), synaptic function (neurogranin), and neuroinflammation (YKL40, GFAP) | 90
  Change from baseline to day 90 in circulating biomarkers of amyloid deposition (Aβ-42, Aβ-40), neuronal/axonal degeneration (t-tau, p-tau, NFL), synaptic function (neurogranin), and neuroinflammation (YKL40, GFAP)
Change in cognition | 90
  Change from baseline to day 90 in cognition, assessed using the Alzheimer's Disease Assessment Scale cognitive subscale 13-item version (ADAS-Cog-13)
Change in instrumental activities of daily living (IADL) | 90
  Change from baseline to day 90 in the Functional Activities Questionnaire (FAQ) score
Change in neuropsychiatric symptoms | 90
  Change from baseline to day 90 in Neuropsychiatric Inventory (NPI) score and 15-item GDS scale score

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital; Neha K Rupeja, MS, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States